CLINICAL TRIAL: NCT06079073
Title: The Effect of Orofacial Myofunctional Therapy With Autofeedback and the Effect of Anatomical and Behavioral Variables on Adherence to Orofacial Myofunctional Therapy in Patients With Mild or Moderate Obstructive Sleep Apnea
Brief Title: The Effect of Orofacial Myofunctional Therapy With Autofeedback on Obstructive Sleep Apnea
Acronym: OMTAOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Oslo Metropolitan University (Other); University of Tartu (Other); Reykjavik University (Other)
Responsible Party: Principal Investigator, Harald Hrubos-Strøm, MD, PhD, senior consultant and head of research group, principal investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/11571
Record Dates: First submitted 2023-08-23; First posted 2023-10-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Block randomization to ensure 40% female participants. Intervention: Access to treatment module in application plus access to OMT therapist. Control: Access to application without treatment module. No scheduled appointments with OMT therapist.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization is conducted at the end of the baseline assessment. Participants in the intervention group is handled by an OMT therapist until outcome assessment by the same postdoc student that did the baseline examination. The postdoc student has not been in contact with any participant during the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application plus treatment module (Experimental): The following exercises are pre-recorded and presented in the treatment module:
  Tongue
  1. Tongue brushing
  2. Tongue sliding
  3. Tongue suction
  4. Tongue down Soft palate
  1. Elevate soft palate and uvula 2. Balloon blow Facial
  1. Put your finger in the oral cavity against your cheek. Pull against your finger with the cheek muscles.
  2. Air pump Exercise adherence is registered in a study application
  Interventions: Behavioral: Orofacial myofunctional therapy with autofeedback
- Application awaiting access to treatment module (No Intervention): Participants receiving a code not unlocking the treatment module will have full access to all other parts of the mobile app. After 90 days, during the outcome evaluation, all participants will receive a new code unlocking the treatment module in order to keep outcome evaluators blinded.

INTERVENTIONS:
Behavioral: Orofacial myofunctional therapy with autofeedback — Participants opening a code unlocking the OMTa treatment module of the application will be given a direct communication link to the PhD students, Diana Hansen (Norway) and Andres Koster (Estonia) and two research co-ordinators. Dr. Hansen and Andres Köster has obtained an Academy of Orofacial Myofunctional Therapy (AOMT) certification diploma. One physical start up session will be scheduled at Ahus and at North Estonia Medical Center. This 60 minute session will be used to instruct participants in OMT exercises and use of the app. All participants will receive a disposable toothbrush and standardized balloons. After that, biweekly video sessions (time 20-30 min) will be scheduled.
  Arms: Application plus treatment module

SUMMARY:
The overall aim of this study is to estimate the effect of orofacial myofunctional therapy (OMT) plus auto-monitoring compared to auto-monitoring alone. Moreover, the investigators aim to identify anatomical and behavioural predictors of OMT adherence

DETAILED DESCRIPTION:
The overall aim will be addressed by reqruiting 100 participants to orofacial myofunctional therapy. 50 will be randomized to immediate treatment after the baseline consultation while 50 will get access to the treatment module after 3 monts of waiting. Outcomes will be assessed by a researcher blinded for the randomization result.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Ahus or the Fertilitas clinic

  * A diagnosis of obstructive sleep apnea according to the current International Classsification of Sleep Disorders (ICSD) version 3 criteria {Berry, 2020, The AASM Manual for the Scoring of Sleep and Associated Events: Rules', Terminology and Technical Specifications', Version 2.6.;, 2014, International classification of sleep disorders', 3rd ed.}, with a respiratory event index (REI) <30.
  * Not previously or currently treated with PAP or MAD
  * Signed informed, written consent.
  * Owning a mobile phone with software compatible for the study application Age ≥18 year.
  * Body mass index <30
  * Ability to breathe through the nose
  * Ability to read and willingness to follow the protocol as described in the written consent form
  * Teeth 5-to 5 should be present or fixed by prosthesis or implants.
  * No botulinium toxin in facial muscles last three months

Exclusion Criteria:

* Failure to fill in at least 70% of days in the electronic sleep diary provided in the mobile app for two weeks.

  * Medical or psychiatric conditions which may interfere with the study protocol in the opinion of the investigator. Examples are acute psychosis, drug abuse and dementia. This will be noted in the study inclusion-exclusion document for each approached candidate for the study. The information will then be discussed in an exlusion committee consisting of dr. Skirbekk, Jagomägi, Dammen and Hrubos-Strøm.
  * Tongue-tie as described below. Participants with mouth opening of <50% with the tip of the tongue at the incisive papilla compared to total mouth opening will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Category "non-binary" possible
Enrollment: 106 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index reduction | 3 months
  Measured by self-applied somnography. The index represents number of apneas or hypopneas per hour from 0/h. Higher values represents more severe disease.

SECONDARY OUTCOMES:
Change in the Epworth Sleepines scale | 3 months
  The scale is a validated tool measuring sleepiness between 0-24. Higher values represent more sleepiness
Orofacial myofunctional therapy adherence | 3 months
  Measured by application registration between 1-3 per day. Three exercises per day is the maximum score
Change in desaturation severity parameter measured by medical device | 3 months
  Measured by photoplethysmography obtained by self-applied somnography. More severity represents more disease.
Change in desaturation duration measured by medical device | 3 months
  Measured by photoplethysmography obtained by self-applied somnography. Longer duration represents more disease.
Change in objective sleep quality | 3 months
  Measured by self-applied somnography. Sleep quality is the ratio between total sleep time and time in bed. A higher ratio is better.
Change in desaturation severity parameter measured by wearable | 3 months
  Measured by photoplethytsmography obtained by Withings Scan Watch. More severity represents more disease.
Change in desaturation duration measured by wearable | 3 months
  Measured by photoplethytsmography obtained by Withings Scan Watch. Longer duration represents more disease.
Change in stroop test | 3 months
  Measured by Flexibility game in application. More correct answers is better
Change in reaction test | 3 months
  Measured by reaction game in application. Shorter reaction time is better
Change in memory test | 3 months
  Measured by memory game in application. Longer sequences memorized is better
Change in perception test | 3 months
  Measured by perception game in application. More correct answers is better.
Change general health status | 3 months
  Measured by a visual analogue scale in the BEAMER questionnaire, two visio analogue scales on general health and 3 items on acceptance and control scored 1-6 respectively.
Changes in the Orofacial Myofunctional Evaluation with Scores | 3 months
  Measured by scorer blinded for randomization. Range 37-103. A lower score represents more dysfunction.
Changes in tongue strength | 3 months
  Objective strength measured by the Iowa Oral Pressure Inventory. A higher score represents more strenght.
Changes in tongue endurance | 3 months
  Objective endurance measured by the Iowa Oral Pressure Inventory. A higher score represents more endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Hrubos-Strøm, PhD, Principal Investigator — University Hospital, Akershus
Locations (2):
- Fertilitas clinic, Tallinn, Estonia
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
Not allowed by Regional Ethical Committee

REFERENCES:
- [Derived] Koster A, Hoang AD, Dashuk A, Vaher H, Sikk K, Jagomagi T. Effects of Web-Based Orofacial Myofunctional Therapy on Hyoid Bone Position in Adults with Mild to Moderate Obstructive Sleep Apnea: Evidence from an Estonian Substudy of a Randomized Controlled Trial. J Clin Med. 2025 Dec 29;15(1):257. doi: 10.3390/jcm15010257. PMID 41517505

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT06079073/Prot_SAP_000.pdf